CLINICAL TRIAL: NCT00029133
Title: Hypothermia During Intracranial Aneurysm Surgery Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01NS038554 (NIH)
Record Dates: First submitted 2002-01-08; First posted 2002-01-09 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-08

CONDITIONS: Aneurysm; Hypothermia; Subarachnoid Hemorrhage
Keywords: aneurysm; hypothermia; subarachnoid intracranial hemorrhage
MeSH Terms: conditions — Aneurysm; Hypothermia; Subarachnoid Hemorrhage

INTERVENTIONS:
Procedure: mild intraoperative hypothermia (33 degrees Celsius)

SUMMARY:
This is a large multi-center, prospective, randomized trial designed to determine whether mild intraoperative hypothermia results in improved neurological outcome in patients with an acute subarachnoid hemorrhage (SAH) who are undergoing an open craniotomy to clip their aneurysms.

DETAILED DESCRIPTION:
The purpose of this trial is to determine whether mild intraoperative body cooling (body temperature = 33 degrees Celsius or 91.4 degrees Fahrenheit) during open neurosurgical craniotomies for aneurysm clipping improves neurological outcome (measured as 3 months after surgery) in patients who have suffered an aneurismal SAH. This may be the only NIH-funded trial to examine the impact of an intraoperative intervention on neurological outcome following any neurosurgical procedure, and is certainly the largest trial of its kind yet undertaken.

Many methods have been proposed to "protect" neurosurgical patients from neurological complications that can occur during and after intracranial vascular procedures. However, no treatment targeted at the intraoperative period has ever been systematically tested. Mild hypothermia was chosen as the treatment to be tested after an extensive review of medical literature and discussions with many anesthesiologists and neurosurgeons expert in the field suggested it was the intervention most likely to be beneficial. Hypothermia is also easily produced in the operating room and most anesthesiologists are familiar with managing mild hypothermia. As a result, the investigators felt that a trial of hypothermia was practical and reasonably safe.

ELIGIBILITY:
* Adult greater than 18 years old
* Non-obese (body mass index less than 35kg/m2)
* Non-pregnant
* World Federation of Neurologic Surgeons preoperative Grade I, II, or III patients with acute SAH and scheduled to undergo open craniotomies for aneurysm clipping within 14 days of a documented SAH.
* There must be no contraindications to cooling (e.g., sickle cell anemia, cryoglobulinemia, or severe Raynaud's disease).
* Patients must also have pre-SAH Rankin disability scores of 0 to 1 (i.e., no serious pre-existing functional disability of any kind), and a perioperative course of Nimodipine (a calcium-channel blocker and the only drug known to improve outcome in patients with SAH) must be planned.
* Each center must have approval from their local Human Subjects Committee to participate in the trial and written informed consent from either the patient, next-of-kin, or legal guardian is required.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2000-02

CONTACTS AND LOCATIONS:
Overall Officials: Michael Todd, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Department of Anesthesia, 6505-5 John Colloton Pavilion, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Bayman EO, Chaloner KM, Hindman BJ, Todd MM; IHAST Investigators. Bayesian methods to determine performance differences and to quantify variability among centers in multi-center trials: the IHAST trial. BMC Med Res Methodol. 2013 Jan 16;13:5. doi: 10.1186/1471-2288-13-5. PMID 23324207